CLINICAL TRIAL: NCT01405599
Title: Evaluation of the Pharmacokinetics, Safety and Tolerability of a Single Dose of Ulimorelin in Subjects With Mild, Moderate and Severe Hepatic Impairment, in Comparison With Healthy Subjects
Brief Title: Evaluation of the Pharmacokinetics of Ulimorelin in Subjects With Hepatic Impairment and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPJ5004-01/2011 (HEP)
Record Dates: First submitted 2011-07-22; First posted 2011-07-29 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Digestive System Disorders
Keywords: Ulimorelin; Hepatic Impairment
MeSH Terms: conditions — Digestive System Diseases | interventions — ulimorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): Healthy subjects
  Interventions: Drug: Ulimorelin
- Severe hepatic impairment (Experimental): CTP class C
  Interventions: Drug: Ulimorelin
- Moderate hepatic impairment (Experimental): CTP class B
  Interventions: Drug: Ulimorelin
- Mild hepatic impairment (Experimental): CTP class A
  Interventions: Drug: Ulimorelin

INTERVENTIONS:
Drug: Ulimorelin — Single dose of 480 micrograms/kg administered as a 30 minute intravenous infusion
  Other Names: TZP101

SUMMARY:
Evaluation of the effect of hepatic impairment on the pharmacokinetics of ulimorelin after a single intravenous (IV) dose in order to identify potential patients at risks in terms of severity of hepatic dysfunction and to determine whether their dosage should be adjusted.

ELIGIBILITY:
Inclusion Criteria:

Main Criteria for Inclusion All Subjects:

* Adult male or female subjects age 18 to 75 years (both inclusive)
* Able to understand and willing to sign an informed consent form (ICF) and able to comply with the study restrictions
* Female subjects must be postmenopausal (for at least 1 year and confirmed by serum follicle-stimulating hormone (FSH) at screening), surgically sterile, practicing true abstinence and/or must be using adequate contraception for the duration of the study (e.g. contraceptive implants, injectables, oral contraceptives, and intra-uterine device and/or barrier methods (condom/occlusive cap with spermicidal foam/gel/film/cream/suppository))
* Females of childbearing potential must have a negative pregnancy test at screening and Day -1
* Weight ≥ 50 kg and ≤ 200 kg
* Body mass index (BMI) ≤ 40.0 kg/m2, where BMI (kg/m2) = Body weight (kg)/Height2 (m2) Inclusion Criteria Hepatic Impairment Subjects (in addition to the criteria for all subjects):
* Documented mild, moderate or severe hepatic impairment defined as either Child-Pugh A, B or C at screening
* Stable hepatic impairment, defined as no clinically significant change in disease status within the last 30 days before screening, as documented by the subject's recent medical history (e.g., no worsening of clinical signs of hepatic impairment and no worsening of total bilirubin or prothrombin time by more than 50%)
* Must be on a stable dose of medication and/or treatment regimen at least 2 weeks before dosing of study medication
* Subjects with a history of substance abuse may be enrolled provided that they have not abused drugs or alcohol for at least 6 months preceding the study Inclusion Criteria for Healthy Subjects (in addition to criteria for all subjects):
* Subjects with normal hepatic function, and liver parameters within normal range unless approved by the Sponsor's Medical Representative
* Subjects not using prescription drugs or non-prescription drugs, including over-the-counter medication, non-routine vitamins and herbal products within 3 weeks prior to dosing of investigational product [use of oral contraceptives, diuretics, noncardioselective beta-blockers, topically applied medication (eye-/nose-drops and creams) and occasional use of metaclopramide, ibuprofen and paracetamol is permitted]. Use of any other medication has to be discussed and agreed before inclusion of the subject with the Medical Monitor and the Sponsor's medical representative

Exclusion Criteria:

Criteria for Exclusion All Subjects:

* Known or suspected allergy to the trial product or related products
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
* Participation in another investigational drug trial within 30 days prior to dosing (or 5 times the half life of the drug if longer)
* Acute illness within 14 days prior to dosing unless mild in severity and approved by the Investigator and Sponsor's medical representative
* History of drug abuse or positive urine drug screen (if not due to concomitant medication) at Screening and/or Day -1
* Ingestion of alcohol and caffeine within 24 hours prior to dosing and for the duration of the study
* Donation of more than 450mL of blood / blood products in the 30 days prior to dosing, and/or blood donation in the 30 days prior to dosing
* Positive result to the screening test for HIV-1 antibodies, HIV-2 antibodies or HIV-1 antigen according to locally used diagnostic testing
* Creatinine clearance <50mL/minute, estimated using serum creatinine with the formula [(140 - age in years) × weight in kg]/[(72 × serum creatinine in mg/dL) × 0.85 for female subjects]
* Consumption of Seville oranges, grapefruit or grapefruit juice, star fruit and exotic fruits from 7 days prior to first dose of study medication and for entire duration of the study
* Clinically significant abnormal haematology, biochemistry, coagulation or urinalysis screening tests, as judged by the Investigator other than the abnormal values expected considering the underlying disease
* Subject with any disease or condition which the Investigator feels would interfere with the trial outcome or compliance except for conditions associated with hepatic impairment in the group of subjects with compromised hepatic function
* Uncontrolled treated/untreated hypertension (systolic blood pressure ≥ 160 mmHg and /or diastolic blood pressure ≥ 105 mmHg)
* Use of prescription or over-the-counter medication that is extensively bound to α1-acid glycoprotein (AAG) which the Investigator or Sponsor feels would interfere with the trial outcome
* History of cancer (judged not to be in full remission) or presence of cancer (except basal cell skin cancer or squamous cell skin cancer) as judged by the Investigator
* Subject who has undergone liver transplantation
* Not able or willing to refrain from smoking during the inpatient period
* Any condition that would make the subject unsuitable for clinical trial participation as judged by the Investigator

Exclusion Criteria Hepatic Impairment Subjects (in addition to criteria for all subjects):

* Any medical or surgical conditions, excluding underlying liver disease, which may significantly interfere with the pharmacokinetics of the study drug
* Fluctuating or rapidly deteriorating hepatic function

Exclusion Criteria for Healthy Subjects (in addition to criteria for all subjects):

* Subjects with clinically significant illness as judged by the Investigator
* Exposure to more than three new chemical entities within 12 months prior to the first dosing day
* Known acute hepatitis with viral, alcoholic, toxic or autoimmunological aetiology within the last 6 months. Positive result to the screening test for Hepatitis B antigen or Hepatitis C antibodies according to locally used diagnostic testing
* Strenuous exercise within 48 hours prior to dosing and for the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cmax of ulimorelin | 15, 30, 45, 60, 75, 90 mins, 2, 4, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 h post-infusion
  To evaluate the pharmacokinetics of ulimorelin in subjects with mild, moderate and severe hepatic impairment compared with subjects who have normal hepatic function following a single dose administration of ulimorelin
AUC of ulimorelin | 15, 30, 45, 60, 75, 90 mins, 2, 4, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 h post-infusion
  To evaluate the pharmacokinetics of ulimorelin in subjects with mild, moderate and severe hepatic impairment compared with subjects who have normal hepatic function following a single dose administration of ulimorelin

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tomas, PhD, Study Director — Norgine
Locations (1):
- Univerzitna nemocnica Bratislava, nem., Bratislava, Slovakia